CLINICAL TRIAL: NCT06619314
Title: A Three-Part Study to Evaluate the Effect of Food, Formulation, and a Proton Pump Inhibitor on the Single-Dose Pharmacokinetics of MK-1084 in Healthy Adult Participants
Brief Title: A Study to Evaluate the Effect of Food, Formulation, and a Proton Pump Inhibitor (PPI) on Calderasib (MK-1084) in Healthy Adult Participants (MK-1084-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1084-003; MK-1084-003 (Other: MSD)
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Calderasib Treatment A (Experimental): Participants will receive calderasib on Day 1 on an empty stomach
  Interventions: Drug: Calderasib
- Calderasib Treatment B (Experimental): Participants will receive calderasib on Day 1 after a high-fat/high-calorie breakfast
  Interventions: Drug: Calderasib
- Calderasib Treatment C (Experimental): Participants will receive calderasib Formulation 1 on Day 1
  Interventions: Drug: Calderasib
- Calderasib Treatment D (Experimental): Participants will receive calderasib Formulation 2 on Day 1
  Interventions: Drug: Calderasib
- Calderasib Treatment E (Experimental): Participants will receive calderasib without a PPI on Day 1
  Interventions: Drug: Calderasib
- Calderasib Treatment F (Experimental): Participants will receive calderasib with a PPI on Day 5
  Interventions: Drug: Calderasib; Drug: PPI

INTERVENTIONS:
Drug: Calderasib — Oral Tablet
  Other Names: MK-1084
Drug: PPI — Oral Capsule
  Arms: Calderasib Treatment F

SUMMARY:
The purpose of this study is to evaluate the effect of food, formulation, and a PPI on the levels of calderasib in a person's body over time.

ELIGIBILITY:
Inclusion Criteria:

* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing.
* Medically healthy with no clinically significant medical history.

Exclusion Criteria:

* Has a history of cancer.
* Has had major surgery and/or donated or lost significant volume of blood.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Food effect: Area Under the Concentration-Time Curve from 0 to Infinity (AUC0-inf) of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the AUC0-inf of calderasib.
Food Effect: Maximum Plasma Concentration (Cmax) of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the Cmax of calderasib.
Formulation Effect: Area Under the Concentration-Time Curve from 0 to the Time of the Last Quantifiable Sample (AUC0-last) of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the AUC0-last of calderasib.
Formulation Effect: AUC0-inf of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the AUC0-inf of calderasib.
Formulation Effect: Area Under the Concentration-Time Curve from 0 to 24 hours (AUC0-24) of Calderasib | At designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24 of calderasib.
Formulation Effect: Cmax of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the Cmax of calderasib.
Formulation Effect: Plasma Concentration at 24 hours (C24) of Calderasib | 24 hours postdose
  Blood samples will be collected to determine the C24 of calderasib.
Formulation Effect: Lag Time (tlag) of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the tlag of calderasib.
Formulation Effect: Time to Maximum Plasma Concentration (Tmax) of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the Tmax of calderasib.
Formulation Effect: Apparent Terminal Half-Life (t1/2) of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the t1/2 of calderasib.
Formulation Effect: Apparent Clearance (CL/F) of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the CL/F of calderasib.
Formulation Effect: Apparent Volume of Distribution During Terminal Phase (Vz/F) of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the Vz/F of calderasib.
Proton Pump Inhibitor (PPI) Effect: AUC0-inf of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the AUC0-inf of calderasib.
PPI Effect: Cmax of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the Cmax of calderasib.

SECONDARY OUTCOMES:
Food Effect: AUC0-last of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the AUC0-last of calderasib.
Food Effect: AUC0-24 of Calderasib | At designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24 of calderasib.
Food Effect: C24 of Calderasib | 24 hours postdose
  Blood samples will be collected to determine the C24 of calderasib.
Food Effect: tlag of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the tlag of calderasib.
Food Effect: Tmax of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the Tmax of calderasib.
Food Effect: t1/2 of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the t1/2 of calderasib.
Food Effect: CL/F of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the CL/F of calderasib.
Food Effect: Vz/F of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the Vz/F of calderasib.
Food Effect: Number of Participants Who Experience a Treatment Emergent Adverse Event (TEAE) | Up to approximately 2 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Food Effect: Number of Participants Who Discontinue Study Treatment Due to a TEAE | Up to approximately 2 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Formulation Effect: Number of Participants Who Experience a TEAE | Up to approximately 2 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Formulation Effect: Number of Participants Who Discontinue Study Treatment Due to a TEAE | Up to approximately 2 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
PPI Effect: AUC0-last of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the AUC0-last of calderasib.
PPI Effect: AUC0-24 of Calderasib | At designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24 of calderasib.
PPI Effect: C24 of Calderasib | 24 hours postdose
  Blood samples will be collected to determine the C24 of calderasib.
PPI Effect: tlag of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the tlag of calderasib.
PPI Effect: Tmax of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the Tmax of calderasib.
PPI Effect: t1/2 of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the t1/2 of calderasib.
PPI Effect: CL/F of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the CL/F of calderasib.
PPI Effect: Vz/F of Calderasib | At designated timepoints (up to 48 hours postdose)
  Blood samples will be collected to determine the Vz/F of calderasib.
PPI Effect: Number of Participants Who Experience a TEAE | Up to approximately 2 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
PPI Effect: Number of Participants Who Discontinue Study Treatment Due to a TEAE | Up to approximately 2 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/